CLINICAL TRIAL: NCT03638856
Title: Comparing Effectiveness of Oral Misoprostal for Cervical Priming in Premenopausal Women Underwent to Diagnostic Hysteroscopy: Double-blind, Randomized Placebo-Controlled Trial
Brief Title: Comparing Effectiveness of Oral Misoprostal for Cervical Priming in Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rjcyto2531
Record Dates: First submitted 2018-06-01; First posted 2018-08-20 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2018-06

CONDITIONS: Abnormal Uterine Bleeding; Chronic Pelvic Pain; Infertility, Female
Keywords: Cervical priming; Diagnosis hysteroscopy; Oral Misoprostal; Premenopause
MeSH Terms: conditions — Metrorrhagia; Infertility, Female | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misoprostal group (Experimental): Patients were added oral Misoprostal 200 mcg 2 tab per oral 3 hour before hysteroscopy
  Interventions: Drug: Misoprostol 200Mcg Tab
- Placebo group (No Intervention): Patients were take placebo 2 tab per oral 3 hour before hysteroscopy

INTERVENTIONS:
Drug: Misoprostol 200Mcg Tab — patient takes 2 tab of 200 mcg of Misoprostal 3 hr before hysteroscopy
  Arms: Misoprostal group

SUMMARY:
Research objective To compare effectiveness of oral Misoprostal for cervical priming in premenopausal women underwent to diagnostic hysteroscopy Research hypothesis: Null hypothesis Effectiveness of oral misoprostal for cervical priming in premenopausal women underwent to diagnostic hysteroscopy is not different from placebo Alternative hypothesis: : Oral Misoprostal for cervical priming in Premenopausal women underwent to diagnostic hysteroscopy is better than placebo

DETAILED DESCRIPTION:
Research design Randomized double-blinded placebo-controlled trial. The investigators who assess the outcomes and the participants do not know Misoprostal group or control group. The patients are given the random concealed envelop which contains Misoprostal or placebo to take before hysteroscopy. Surgeon and the investigator whom assess patients do not know group allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal women
2. Patients have following indication for diagnosis hysteroscopy

   * Abnormal uterine bleeding
   * Unexplained infertility
   * Recurrent pregnancy loss
   * Chronic pelvic pain
   * Late postpartum hemorrhage
3. Patients provided written informed consent

Exclusion Criteria:

1. Postmenopausal women
2. Patients who have contraindication for Misoprostal as following

   * Allergic to Misoprostal
   * Medical illnesses such as cardiovascular diseases, Asthma, Renal disease
3. Patients who have contraindication for Hysteroscopoy as following

   * Pregnant women
   * Pelvic inflammatory disease
   * Infection at cervix and vagina
   * Cervical cancer

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — need to evaluation of cervical priming
Enrollment: 17 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
initial cervical diameter | 1 year
  The initial hedgar dilator number which can easily insert through cervix

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand